CLINICAL TRIAL: NCT04390100
Title: Palatal Wound Healing Evaluation After Application of Platelet Rich Fibrin Versus 0.2% Hyaluronic Acid Dressings (Randomized Controlled Clinical Trial)
Brief Title: Palatal Wound Healing Evaluation After Application of Platelet Rich Fibrin Versus 0.2% Hyaluronic Acid Dressings
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nourhan Alaa el din Akl, principal investigator(teaching assistant), Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 566
Record Dates: First submitted 2020-05-09; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Free Gingival Graft
MeSH Terms: interventions — Hyaluronic Acid; Gels; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Intervention Model Description: 3 groups each receiving a different type of intervention
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRF (Active Comparator): PRF membrane is placed in the area where the free gingival graft was taken from the palate
  Interventions: Other: Platelet rich fibrin
- hyaluronic acid (Active Comparator): hyaluronic acid gel is placed in the area where the free gingival graft was taken from the palate and the patient is instructed to place the gel 3 times per day
  Interventions: Drug: hyaluronic acid (Gengiegel 0.2% oral gel )
- Gel foam (Active Comparator): Gel foam is placed in the area where the free gingival graft was taken from the palate
  Interventions: Other: Gel foam

INTERVENTIONS:
Drug: hyaluronic acid (Gengiegel 0.2% oral gel ) — coverage of the free gingival graft area in the palate
  Other Names: Platelet rich fibrin (PRF)
  Arms: hyaluronic acid
Other: Platelet rich fibrin — coverage of the free gingival graft area in the palate
  Other Names: PRF
  Arms: PRF
Other: Gel foam — coverage of the free gingival graft area in the palate
  Arms: Gel foam

SUMMARY:
Free gingival graft (FGG) was first proposed by Bjorn 1963 and Nabers 1966. FGG is indicated to correct mucogingival problems such as inadequate or lack of attached gingiva and gingival recession. The most frequent donor site for free gingival graft is the palate

Although, great concern has been given to the recipient sites by using different techniques as suturing, tissue adhesives and special dressings, a little attention was given to protect the donor sites after free gingival graft harvesting. The palatal donor site heal by secondary intention, it could take around 2 to 4 weeks depending on the width and thickness of the tissue removed.The common clinical events that occurs following FGG procedure are patient's discomfort, pain and bleeding at the donor site.

DETAILED DESCRIPTION:
In an attempt to protect the plate (donor site) so that it could help in decreasing the patient's post operative pain, Farnoush suggested variant clinical techniques. One of these techniques was interproximal wire ligation by placing a stainless steel wire anchored on the teeth stabilizing the periodontal dressing. He also suggested using a modified Hawley appliance which would act as a palatal stent protecting the palate to help in healing.

After periodontal surgeries, the donor site (palate) has to be protected from the external environment by many dressing materials. Conventional periodontal dressings provide an inert barrier that help healing by preventing the external insults on the wound area. However, these dressings do not affect the cellular behavior and do not display a role in the biological events that happen during wound healing.

Platelet-rich fibrin (PRF) is a simple procedure where patient's own blood is collected and centrifuged. PRF clot forms a strong fibrin matrix that can be compressed to form a membrane. PRF membrane consists of a fibrin 3D mesh polymerized in a specific structure that incorporates platelets, leukocytes, growth factors; and the circulating stem cells.PRF membrane enhance angiogenesis, immunity and wound epithelialisation. Thus, based on such findings the PRF membrane can be used as a palatal dressing

PRF membrane enhances the healing of the donor site (palate).According to Shakir et al., complete epithelialisation of the palatal donor site was reached by 18th day after FGG in the groups where PRF membranes was placed with less pain scores on the 2nd and 7th day than the control group. Therefore PRF membranes showed higher capabilities of the donor site healing stimulation.

Hyaluronic acid (HA) is a high molecular weight, non-sulphated polysaccharide component of the family of the glycosaminoglycanes,it is present in various body fluids such as synovial fluid, serum, saliva and gingival crevicular fluid. In addition, it represents an important component of the extracellular matrix of skin, connective tissue, synovial joints and other tissues. HA is identified in all periodontal tissues, being prominent in the non-mineralized tissues such as gingiva and periodontal ligament, and in low quantities in mineralized tissues such as cementum and alveolar bone.

Hyaluronic acid has been suggested as monotherapy or as an adjunct to non-surgical and/or surgical periodontal treatment to reduce inflammation and promote wound healing. Hyaluronic acid can be used to accelerate the palatal wound healing at the donor site after free gingival graft surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients who are indicated for soft tissue augmentation with free gingival graft for mucogingival surgery or for implant therapy
* Good patient compliance with the plaque control instructions following initial therapy.

Exclusion Criteria:

* Presence of systemic diseases which could influence the outcome of the therapy
* Smoker patients.
* Pregnant females
* Vulnerable group of patients (prisoners ,handicapped, decisionally impaired individuals)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
visual analogue scale(VAS) | one month
  evaluate of the pain at 3,7,14,21 and 30 with score staring from 0 (minimal pain) to 10(maximum pain) after the application of Platelet rich fibrin and hyaluronic acid and gel foam as a palatal dressing after harvesting a free gingival graft from the palate (donor site)

SECONDARY OUTCOMES:
assessment of healing using the healing index scale by Landry et al1984 | one month
  evaluate the palatal healing at 7,14 21 and 30 days with scale starting from (1 for very poor healing and 5 excellent healing) following free gingival graft harvesting using Platelet rich fibrin and hyaluronic acid.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed abdel aziz hassan, Associate Professor, Study Director — faculty of dentistry ain shams university
Locations (1):
- Faculty of Dentistry ,Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
sharing of the study methodology and the clinical results
Supporting Information: Study Protocol, CSR
Time Frame: the data will be available for a year from it's submission date

DOCUMENTS (1):
  • Study Protocol (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT04390100/Prot_000.pdf